CLINICAL TRIAL: NCT03381040
Title: Predictive Algorithm for Product Selection in the Management of Mid Facial Volume Correction: Part I - A Pilot Validation of Patient Strata
Brief Title: Midfacial Product Selection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-01-001G
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Facial Volume Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Poor structural support/volume (atrophy of soft tissues, leading to loss of projection) with adequate skin envelope (normal or thick skin). Treated with Restylane Lyft.
  Interventions: Device: Restylane Lyft
- Group B (Active Comparator): Poor structural support/volume (atrophy of soft tissues, leading to loss of projection) with poor skin envelope (thin skin). Treated with Restylane Volyme.
  Interventions: Device: Restylane Volyme

INTERVENTIONS:
Device: Restylane Lyft — Restylane® Lyft is a sterile gel of hyaluronic acid with lidocaine generated by Streptococcus species of bacteria, chemically cross-linked with BDDE (the cross linker), stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL. Lyft is intended to be used for facial tissue augmentation. It is recommended that the product be used for shaping the contours of the face and the correction of folds using the co-packed needles. Given the very high lift capacity of Lyft, it is often used when the skin envelope is normal or thicker than normal, as the contours of the product may be palpable in the presence of thin skin.
  Arms: Group A
Device: Restylane Volyme — Restylane® Volyme is a sterile, biodegradable, viscoelastic, non-pyrogenic, clear, colorless, and homogeneous soft hyaluronic acid gel with a high lifting capacity. Volyme is intended for injection into the supraperiostic zone or subcutis to augment the volume of the cheeks.
  Given Volyme's viscoelastic and lifting capacities, it is best used when there is significant loss of volume and a thin skin envelope.
  Arms: Group B

SUMMARY:
This study seeks to determine whether patients pursuing injectable treatments for facial volume loss and/or contour deficiency can be separated into strata based on characteristics such as skin envelope and subcutaneous tissue quantity in the zygomatic, submalar and anteromedial cheek regions in order to guide the clinician in making the ideal product choice (i.e., Restylane Volyme vs Lyft)?

DETAILED DESCRIPTION:
With age, loss of facial fat and hollowing of the cheeks can result in a "sinking" appearance in the mid-face. Augmentation and contouring of the area can be corrected using dermal fillers such as Restylane.

Currently, product choice and amount of volume used for injectable procedures varies between physicians as there is no standard for treatment. Individual assessment based on the attending physician's preference and experience determines final product selection and technique. An algorithm is needed to standardize best practices between physicians and clinics and to better regulate the use of dermal fillers in facial plastic surgery.

Therefore, the purpose of this study is to is to develop an algorithm to decide on which product (i.e., Restylane Volyme or Lyft) to use in the cheek area based on subject characteristics such as age, skin quality, subcutaneous fat quantity and positioning, and bony structure.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of consent, women between the ages of 30 and 75 years old;
2. Patients with established mid-face/cheek hollowing;
3. Patients with a MMVS score of 2 or 3 at baseline;
4. Accepted the obligation not to receive any other facial procedures through the 4-month follow-up;
5. Understood and accepted the obligation and would be logistically able to appear for all scheduled follow-up visits;
6. No previous facial fillers for a period of 12 months prior to this study;
7. No previous facial fillers in the mid-face for 18 months prior to this study;
8. Capable of providing informed consent.

Exclusion Criteria:

1. Current Pregnancy or lactation [sexually active women of childbearing age must agree to use medically acceptable methods of contraception for the duration of this study (e.g., oral contraceptives, condoms, intrauterine device, shot/injection, patch)].;
2. Hypersensitivity to Restylane products, hyaluronic acid filler or amide local anesthetics;
3. Patients presenting with porphyria;
4. Inability to comply with follow-up and abstain from facial injections during the study period;
5. Heavy smokers, classified as smoking more than 12 cigarettes per day;
6. History of severe or multiple allergies manifested by anaphylaxis;
7. Previous tissue revitalization therapy in the treatment area within 6 months before treatment with laser or light, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling, or dermabrasion;
8. Previous surgery including aesthetic facial surgical therapy or liposuction, piercing, or tattoos in the treatment area;
9. History or presence of any disease or lesion near or at the treatment area, including inflammation, active or chronic infection, including in the mouth, dentals, head and neck region;
10. Facial psoriasis, eczema, acne, rosacea, perioral dermatitis and herpes zoster;
11. Scars or deformities;
12. Cancer or precancer, e.g. actinic keratosis;
13. History of radiation therapy to the treatment area;
14. History of bleeding disorders or treatment with thrombolytics, anticoagulants, or inhibitors of platelet aggregation (e.g. Aspirin or other non-steroid anti-inflammatory drugs [NSAIDs]), within 2 weeks before treatment;
15. Patients using immunosuppressants;
16. Patients with a tendency to form hypertrophic scars or any other healing disorders;
17. Patients with known hypersensitivity to lidocaine or agents structurally related to amide type local anaesthetics (e.g., certain anti-arrhythmics);
18. Patients administered dental block or topical administration of lidocaine;
19. Patients with epilepsy, impaired cardiac conduction, severely impaired hepatic function or severe renal dysfunction.
20. Skin thickness between 1.2mm and 1.49mm (as determined by ultrasound).

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Comparison of two Restylane products to treat mid-face/cheek deformities. | Baseline and Week 16.
  Investigators will evaluate whether a difference in physician assessed efficacy as per the standardized photos between two Restylane products at 16 weeks (visit 5) in comparison to baseline (visit 1) using the GAIS scale.

SECONDARY OUTCOMES:
Standardized Imagery for the Improvement of Mid-face Hollowing | Baseline to week 8
  Investigators will evaluate whether an aesthetic change in mid-face contour is observed at visit 3 (4 weeks), and visit 4 (8 weeks) compared to Baseline. The change in mid-face shape will be assessed using the standardized photographs.
Patient satisfaction questionnaire | Baseline to 16 weeks
  Patients will rate their overall satisfaction with treatment results using the patient satisfaction questionnaire at visits 2, 3, 4 and 5. The questionnaire is a 5-point scale comprising 'extremely satisfied', 'satisfied', 'slightly satisfied', 'dissatisfied', and 'extremely satisfied'.
Global aesthetic improvement scale | Baseline to 16 weeks
  Physicians will rate the overall improvement since injection using the Global Aesthetic Improvement Scale at visits 2, 3, 4 and 5. The scale is a 5-point scale comprising 'very much improved', 'much improved', 'improved', 'no change', and 'worse'.
Medicis Mid-face Volume Scale | Baseline to 16 weeks
  At visits 2, 3, 4 and 5, a blinded reviewer will rate each patient's hemiface using the MMVS. The MMVS is a four-point scale that measures the amount of mid-face volume loss comprising of "fairly full", "mild loss", "moderate loss" and "substantial loss". MMVS response rate, defined as the percentage of subjects with at least a 1-grade improvement in MMVS from Baseline up to Week 16 after treatment, will be used in the analyses.
Standardized Ultrasonography Images | Baseline to 16 weeks
  Ultrasound images will be taken before and after injections at the Baseline visit, and all subsequent follow up visits. At Visit 1, the images will be used to determine skin thickness and ascertain the site (e.g., dermis, subcutaneous region) of filler injected into the soft tissue of the face. At follow up visits, ultrasound images will be used to delineate whether the amount of filler has decreased between visits. The analyses of the sonographic characteristics of the fillers will allow for optimization of treatment results.

OTHER OUTCOMES:
Adverse events | Baseline to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Victoria Park Clinical Research Centre, Westmount, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No